CLINICAL TRIAL: NCT02489734
Title: Association Between Post Extubation Delirium and Pre-extubation End-tidal Sevoflurane Concentration in Children
Brief Title: Post Extubation Delirium and End-tidal Sevoflurane Concentration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EDETSC
Record Dates: First submitted 2015-06-16; First posted 2015-07-03 (Estimated); Results first posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2020-08

CONDITIONS: Delirium on Emergence
Keywords: sevoflurane; emergence delirium; preschool
MeSH Terms: conditions — Emergence Delirium | interventions — Sevoflurane

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- low concentration (LC) (Experimental): low concentration group
  Interventions: Drug: sevoflurane
- high concentration (HC) (Experimental): high concentration group
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: sevoflurane — extubation when end-tidal concentration of sevoflurane < 0.5%
  Arms: low concentration (LC)
Drug: Sevoflurane — extubation when end-tidal concentration of sevoflurane >= 0.5%
  Arms: high concentration (HC)

SUMMARY:
The purpose of this study is to determine whether the incidence of emergence delirium will be reduced when end-tidal concentration of sevoflurane decreases.

DETAILED DESCRIPTION:
Sevoflurane induction and maintenance were selected. Intubation was performed after lidocaine spray on vocal cord. After that, an effective caudal or brachial plexus block was performed. End-tidal concentration of sevoflurane was maintained at 2.5%. Spontaneous respiratory was maintained. Sevoflurane was stopped after the end of surgery. Patients were randomly assigned to 2 groups: high concentration group (Group HC, end-tidal concentration of sevoflurane when extubating >=0.5%) and low concentration group (Group LC, end-tidal concentration of sevoflurane when extubating <0.5%). Patients in Group LC were extubated when they coughed or purposeful movement appeared. The patients whose end-tidal concentration of sevoflurane >= 0.5% were excluded. Patients in Group HC were extubated when any of the criteria was met: 1.the patient coughed or purposeful movement appeared 2.end-tidal concentration of sevoflurane decreased to 0.5%. A trained nurse (blind to groups) recorded PAEDs scores in PACU.

ELIGIBILITY:
Inclusion Criteria:

* Age 2-7 years
* ASA I - II
* Estimated surgery time < 2 hours
* Sevoflurane induction and maintenance along with caudal block or Axillary Block

Exclusion Criteria:

* Craniofacial anomalies
* Difficult exposure of the vocal cordS
* Obesity
* Asthma
* Invalid caudal block or axillary block

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 109 (Actual)
Dates: Start 2015-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xuan Wang, Principal Investigator — Children's Hospital of Fudan University

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From July 2015 to September 2015, 135 patients were assessed for eligibility in Children's Hospital of Fudan University.
Pre-assignment Details: Of 135 patients assessed for eligibility, 26 patients were excluded because they did not meet the inclusion criteria or declined to participate in the study.
Period: Overall Study
Arm/Group | Low Concentration (LC) | High Concentration (HC)
Started | 56 | 53
Completed | 39 | 53
Not Completed | 17 | 0

BASELINE CHARACTERISTICS:
Groups:
- Low Concentration (LC): In the LC group, the trachea was extubated as soon as cough or purposeful movement appeared when end-tidal sevoflurane concentration was less than 0.5%. Patients were excluded in this group if cough or purposeful movement appeared when end-tidal sevoflurane concentration was more than 0.5%.
- High Concentration (HC): In the HC group, when end-tidal sevoflurane concentration was more than 0.5%, the trachea was extubated as soon as cough or purposeful movement appeared. If there was still no cough or purposeful movement when end-tidal sevoflurane concentration had decreased to 0.5%, the trachea was extubated at this concentration.
- Total: Total of all reporting groups
Arm/Group | Low Concentration (LC) | High Concentration (HC) | Total
Number analyzed (Participants) | 39 | 53 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.4 (1.4) | 3.9 (1.5) | 3.7 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 31 | 43 | 74
Weight [Mean (Standard Deviation); unit: kg] — obtained from the hospital information system
  kg | 18.2 (4.4) | 19.5 (4.9) | 18.9 (4.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Emergence Delirium (ED)
Description: The primary outcome was the number of participants with emergence delirium (ED) according to the peak PAED score measured by Pediatric Anesthesia Emergence Delirium Scale. All PAED (Pediatric Anesthesia Emergence Delirium scale) scores were assessed by a dedicated nurse who was blinded to the random assignment of patients to group. PAED scores were assessed on awakening (defined as reactive to verbal command or opening of eyes or crying in response to slight touch) and then every 5 minutes for 30 minutes. If the PAED score was ≥ 16, propofol 1 mg.kg-1 was administrated. After administration of propofol, PAED scores were no longer assessed. The peak (highest) PAED score for each patient was analyzed. ED was defined as a peak PAED score >12. Higher score of PAED means a worse outcome.
Time Frame: within 30 minutes after awakening
Measure: Count of Participants; unit: Participants
Arm/Group | Low Concentration (LC) | High Concentration (HC)
Number analyzed (Participants) | 39 | 53
Participants | 5 | 23
Statistical Analysis 1: Comparison: Low Concentration (LC) vs High Concentration (HC); Test type: Superiority; p = 0.003, Chi-squared; Relative risk (RR) = 3.4, 95% CI 2-sided [1.4 to 8.1]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed and recorded during the PACU, an average of 1 hour.
Description: In the PACU, any adverse events such as hypoxemia (defined as SpO2 <92%), laryngospasm (defined as inability to ventilate despite maneuvers to relieve airway obstruction), bronchospasm (defined as wheezing on auscultation), respiratory obstruction (defined as chin lift, oral airway, or reintubation needed to avoid hypoxemia), or postoperative nausea and vomiting (PONV) were recorded by the same nurse.
Arm/Group | Low Concentration (LC) | High Concentration (HC)
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/53
Other Adverse Events (participants affected / at risk) | 3/39 | 5/53
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Concentration (LC) (N=39) | High Concentration (HC) (N=53)
respiratory obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 3 — Respiratory obstruction was defined as chin lift, oral airway, or reintubation needed to avoid hypoxemia.
postoperative nausea and vomiting (Gastrointestinal disorders) | 3 | 2
hypoxemia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 — defined as SpO2 <92%
laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 — defined as inability to ventilate despite maneuvers to relieve airway obstruction
bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 — defined as wheezing on auscultation

LIMITATIONS AND CAVEATS:
First, the patients might have experienced pain in the PACU. However, distinguishing ED from pain in the PACU could be difficult.

Second, we did not observe the duration of each case of ED.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes